CLINICAL TRIAL: NCT05018546
Title: Safety and Efficacy of Gravity Irrigation Versus Pressure Irrigation in Retrograde Intrarenal Surgery (RIRS): A Randomized Controlled Trial
Brief Title: Safety and Efficacy of Different Irrigation System in Retrograde Intrarenal Surgery
Acronym: RIRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Collaborators: Nepal Health Research Council (Other Government)
Responsible Party: Principal Investigator, Dr Purushottam Parajuli, Principal Investigator, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 21/(6-11)/E2/077/078
Record Dates: First submitted 2021-07-13; First posted 2021-08-24 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Urinary Tract Infections; Ureteric Injury; Sepsis
MeSH Terms: conditions — Urinary Tract Infections; Sepsis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gravity Irrigation (Experimental): RIRS under Gravity irrigation
  Interventions: Procedure: Irrigation force
- Pressure Irrigation (Experimental): RIRS under Pressure irrigation.
  Interventions: Procedure: Irrigation force

INTERVENTIONS:
Procedure: Irrigation force — RIRS with different irrigation force

SUMMARY:
Urolithiasis is one of the most prevalent urological diseases affecting general population across the world. The available treatment modalities for renal stones are Shock wave lithotripsy (SWL), Percutaneous Nephrolithotomy (PNL), and Retrograde Intrarenal Surgery (RIRS). Irrigation for RIRS is the critical component for the success of procedure. To avoid detrimental effects of high pressure, intra-renal pressure (IRP) has to be lower. Different studies have shown that high irrigation pressure raises intra-renal pressure leading to pyelo-venous and pyelo-lymphatic reflux which can lead to sepsis and septic shock. Comparative study of different irrigation pressure during RIRS is lacking.

This is randomized controlled trial conducted in Department of Urology and Renal Transplant Surgery for duration of one year. Objective of the study is to compare safety and efficacy of gravity irrigation versus pressure irrigation. Patients with symptomatic kidney stones: non lower pole stones <2cm, lower pole stones <1cm and lower pole stones 1-2 cm in whom PCNL is contraindicated will be enrolled in study with informed consent. Retrograde intrarenal surgery will be performed as standard procedure and Ho:YAG laser will be used to fragment stones.

Stone free rate at postoperative day 1 and after 1 month will be monitored through X-ray KUB. Maximum irrigation pressure, duration of surgery, stone size, density, location, intraoperative and postoperative complications as classified by Clavien-Dindo will be noted for all patients. Data will be appropriately analyzed and statistical tests applied as necessary.

DETAILED DESCRIPTION:
Introduction Urolithiasis is one of the most prevalent urological diseases affecting general population across the world. The worldwide prevalence ranges from 7%- 13% in North America, 5%-9% in Europe, and 1%-5% in Asia.1 West Asia, Southeast Asia, South Asia as well as several developed countries, including South Korea and Japan, have been categorized into stone forming belt countries with prevalence ranging from 5% to 19.1%. Increasing incidence of stone disease is linked with modern life style, food habits, climate as well as increasing use of imaging (computed tomography or ultrasonography)2,3,4 Renal stones constitute about 80% of total urolithiasis. Shock wave lithotripsy(SWL), Percutaneous Nephrolithotomy(PNL), and Retrograde Intrarenal Surgery (RIRS) are available treatment modality for renal stones. According to European Association of Urology (EAU) 2020 Guidelines, when active treatment of renal stones of size <10 mm is indicated, primary treatment modality is either SWL or RIRS. For stones of size > 20 mm, PNL is first line of treatment, however if it is contraindicated then RIRS or SWL can be used. Stones of size 10-20 mm in non-lower pole calyx can be dealt with SWL or Endourology (PNL or RIRS). Lower pole calyx stones of 10-20 mm with unfavorable factors like steep infundibulo-pelvic angle, long calyx, long skin to stone distance, narrow infundibulum and shock wave resistant stones need to be treated with endourology (PNL or RIRS). However, favorable lower pole calyx stones of size 10-20 mm are recommended for SWL or Endourology.5According to AUA guidelines6, in symptomatic patients with a total non-lower pole renal stone burden ≤ 20 mm, SWL or RIRS can be offered. Patients with a total renal stone burden > 20 mm, PNL are the first line therapy. For patients with < 10 mm lower pole renal stones, SWL or RIRS is first line treatment. Patients shouldn't be offered SWL as first line therapy to lower pole stones >10 mm. Patients with lower pole stones >10mm in size need to be explained that PNL has a higher stone free rate but greater morbidity.

RIRS is occasionally associated with severe infectious complications.14 Reasons commonly attributed to it are high intra-pelvic pressure, obstruction, infected urine and stone, break in sterility of procedure etc. Ureteral Access Sheath (UAS) is one of the measure used to decrease intra-pelvic pressure during stone fragmentation.13 Irrigation for RIRS is the critical component for the success of procedure. For better vision during procedure, irrigation pressure (IP) and irrigation flow (IF) needs to be increased. To avoid detrimental effects of high pressure, intra-renal pressure (IRP) has to be lower than 22 mmHg (30 cm of water (H2O))7. High pressure irrigation raises intrarenal pressure leading to pyelo-venous and pyelo-lymphatic reflux which can lead to sepsis, septic shock, bleeding, infundibular rupture.

Some studies have estimated that at an IP of ≤ 100 cm H2O (73 mmHg), IRPs remain lower than 30 cm H2O if Ureteric Access Sheath (UAS) bigger than 10/12 F is utilized. An IP of 200 cm H2O (146 mmHg) may offer high irrigation flows but could result in IRPs > 40 cm H2O8,9. During forced irrigation and stone fragmentation, IRP can rise upto 300mmHg for short interval.15 Omar M. et al in another similar endourological procedure, PCNL which showed High Irrigation Pressure (272 cm H2O) to be associated with a higher risk of SIRS (46%) compared to low Irrigation Pressure (108.8 cm H2O) risk of 11%.10 Gravity irrigation at 100 cm of H2O (73 mmHg), exerts IRP lower than 30 cm of H2O, however in pressure irrigation IRP increases significantly higher. In this study Investigators want to compare between two groups in terms of safety and efficacy.

Rationale and Justification of study Irrigation is required in RIRS for better vision and smooth performance of surgery. However, high IP during RIRS is implicated for infective complications. Comparative study of different pressures for irrigation during RIRS is lacking. Investigators would like to study the safety and efficacy of gravity irrigation versus pressure irrigation in RIRS.

Objectives

General objectives To study the safety and efficacy of gravity irrigation versus pressure irrigation in RIRS Specific objectives

1. To study the demographic pattern of patients undergoing RIRS
2. To compare complications rate of gravity irrigation versus pressure irrigation in RIRS
3. To identify the stone clearance of gravity irrigation versus pressure irrigation in RIRS
4. To compare duration of stone fragmentation of gravity irrigation versus pressure irrigation in RIRS

   Research question Which irrigation system is safe and efficacious: gravity or pressure irrigation? Research Hypothesis Null hypothesis There is no difference in terms of safety (complications and length of hospital stay) and efficacy (stone free rate and fragmentation time) between gravity and pressure irrigation in RIRS.

   Alternative hypothesis There is difference in terms of safety and efficacy between gravity and pressure irrigation in RIRS.

   Research design and Methodology

   Research method- Quantitative

   Types of study- Prospective Randomized Controlled Trial

   Study population- Patients undergoing RIRS surgery for renal calculi and who give consent for study

   Study site - Department of Urology and Renal Transplant Surgery

   Sampling method -Random sampling

   Sample size- Sample size calculation

   N= 2 * { (Z 1-α + Z 1-β) / (d-δ)}2 *p* (1-p)

   Basis for sample calculation is study by Omar M et al in another similar endo-urological procedure, PCNL which showed High Irrigation Pressure (272 cm H2O) to be associated with a higher risk of SIRS (46%) compared to low (108.8 cm H2O) Irrigation Pressure 11%).10

   Expected time and duration of the study- 1 year

   Tools and techniques for data collection

   Data collection will be done using preformed proforma and entered in windows excel. Patient's demographic profile, stone characteristics and pelvi-calyceal anatomy will be recorded. Categorical variables will be expressed as proportions (%) and continuous variables expressed as Mean ± Standard Deviation(SD). Chi-square test will be used for categorical data and Mann-Whitney U test or student's t test will be applied for continuous variables as appropriate.

   Management protocol of patients

   Patients with symptomatic renal calculi fulfilling inclusion criteria, will be considered for RIRS. Pre-operative workup of patients includes Complete blood count, Renal function test, Chest X ray, Electrocardiogram (ECG), Urine routine and microscopy, Urine culture and sensitivity. Imaging work-up includes X-ray Kidney Ureter and Bladder (KUB), Ultrasonography Abdomen and Pelvis and Computed Tomography (CT) Urography. Pre-operatively R.I.R.S. scoring system is used to predict stone free rate.11 Patient planned for surgery needs sterile urine. If patient has indwelling tube/catheter and urine culture shows colonized organism, then patient will be treated with sensitive antibiotics for at least 3 doses. Informed written consent will be taken from patient and patient information sheet (PIS) will be given. Patient will be randomized to two groups: gravity irrigation group and pressure irrigation group in 1:1 ratio through computer generated random numbers. Even numbers will be assigned to gravity irrigation group and odd numbers to pressure irrigation group. Patient will get prophylactic antibiotic at the time of induction with single dose of ceftriaxone 1gm IV and amikacin 750 mg IV or sensitive antibiotics will be continued.

   Patient will be placed in lithotomy position and rigid cystoscopy (19 Fr sheath and 30 scope) will done. Guidewire (Terumo 0.035 inch) will be parked into renal pelvis and ureteric access sheath 9.5/11.5 Fr (Cook Medical, Bloomington) will be placed reaching just proximal ureter under fluoroscopy. Flexible ureteroscopy will be done with Karl Storz FLEX X2S connected to irrigation system consisting of intravenous infusion set (JMS® Singapore PTE LTD, Singapore) connected to 1 Liter (L) normal saline compressible plastic bottle (Aculife®, Aculife Healthcare Pvt. Ltd, Gujarat, India) placed at height of 100 cm from patient's symphysis pubis. In Gravity irrigation group, RIRS surgery will be done with 1 L normal saline bottle placed at 100 cm from patient's symphysis pubis. In case of poor vision and procedure can't be completed with gravity irrigation, pressure irrigation will be used and this conversion will be mentioned in proforma. In pressure irrigation group, Irrigation pressure will be given by arterial line pressure bag and will be started from 80 mmHg and subsequently increased by 10 mmHg as required and peak irrigation pressure required will be noted.

   Stones will be dusted and fragmented with laser energy (LithoDK30, Holmium 2.1 micrometer, Quanta System, Milan, Italy). Duration of surgery along with stone fragmentation time will be noted. After the procedure, DJ stent will be placed and removed after 2 weeks.

   Stone clearance will be confirmed fluoroscopically at the completion of surgery, Post operative day one (POD1) and Post operative month one (POM1) with X-ray KUB and USG abdomen and pelvis. If patient requires more than one stage procedure, it will be mentioned. Patient's post-operative course will be monitored and any complications will be noted. For rapid identification of sepsis, quick Sequential Organ Failure Assessment (qSOFA) score will be used: respiratory rate of 22/min or greater, altered mentation, or systolic blood pressure of 100 mmHg or less. qSOFA score more than two alerts to evaluate for sepsis and septic shock. Double J (DJ) stent will be placed for 2 weeks unless its removal required because of fever. Post-operative complications will be recorded as per classification described by Clavien-Dindo.12

   Process of data Analysis Data collected in Proforma will be entered in Windows Excel. Comparative analysis will be done between gravity irrigation versus pressure irrigation.

   CONSORT Flow Diagram

   Plan for data management and statistical analysis

   Data collection will be done in proforma and will be entered in Windows Excel. Patient's demographic profile, stone characteristics and pelvi-calyceal anatomy will be recorded. Categorical variables will be expressed as proportions (%) and continuous variables expressed as Mean ± SD. Chi-square test will be used for categorical data and Mann-Whitney U test or student's t test will be applied for continuous variables as appropriate. P value of <0.05 will be considered significant.

   Biases and Limitations of the study

   During procedure, vision is subjective and depends on surgeon's assessment and may require high pressure to obtain optimum vision. Surgeon's patience is required to wait till vision becomes clear. Size of stone, type and volume of stone, use of ureteric access sheath, past history of DJ stent placement, past history of endourological procedure as well as patient's comorbidities like diabetes mellitus, immunocompromised status can be confounding factors for longer duration of surgery, complications and stone clearance rate.

   Safety considerations During evaluation and treatment of patient, safety and care of patient will be taken. No unnecessary intervention or medication will be given to patient apart from what is mentioned in our study and current best practice for management of renal stones.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic renal stone <2cm in renal pelvis, upper, middle pole calyx or pelviureteric junction
2. Lower pole stone < 1cm
3. Lower pole stone 1-2 cm when PCNL is contraindicated or not patient's preference
4. Asymptomatic stone of size >15 mm

Exclusion Criteria:

1. Age below 18 yrs
2. Stone >2 cm
3. Ureteric stone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
INFECTION | within 30 days
  urinary tract infection, sepsis, septic shock
stone clearance | within 30 days
  stone clearance assessed with x-ray and USG abdomen

CONTACTS AND LOCATIONS:
Overall Officials: Purushottam Parajuli, MBBS,MS, Principal Investigator — Tribhuvan University Teaching Hospital
Locations (1):
- Tribhuvan University Teaching Hospital, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Yes
study protocol, statistical analysis plan, Informed consent form will be shared. Result and Master chart will also be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 5 years
Access Criteria: Government research body, Journal editors, authors who request will be provided